CLINICAL TRIAL: NCT00573781
Title: Systems Biology Approach to Understand Dietary Modulation of Gene Expression and Metabolic Pathways in Subjects With Abnormal Glucose Metabolism (Sysdimet)
Brief Title: Dietary Modulation of Gene Expression and Metabolic Pathways in Glucose Metabolism
Acronym: Sysdimet
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Marjukka Kolehmainen (Other)
Collaborators: VTT Technical Research Centre, Finland (Other); Wageningen University (Other)
Responsible Party: Sponsor-Investigator, Marjukka Kolehmainen, Senior scientist, University of Eastern Finland
Organization: University of Eastern Finland (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 56/2007; 117844 by Finnish Academy
Record Dates: First submitted 2007-12-13; First posted 2007-12-14 (Estimated); Last update posted 2012-04-17 (Estimated); Status verified 2012-04

CONDITIONS: Metabolic Syndrome; Obesity; Impaired Glucose Tolerance; Impaired Fasting Glucose
Keywords: Systems biology; Nutrigenomics; Metabolomics; Gene expression; Fat tissue; Peripheral mononuclear cells; Gene clusters; Gene expression profiles; Personal diets; Metabolic syndrome; Type 2 Diabetes; Atherosclerosis
MeSH Terms: conditions — Metabolic Syndrome; Obesity; Glucose Intolerance; Diabetes Mellitus, Type 2; Atherosclerosis | interventions — Diet; Fruit; In Situ Hybridization, Fluorescence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Experimental): Diet with increased intake of rye bread, berries and fish
  Interventions: Dietary Supplement: Diet with increased intake of rye bread, berries and fish
- B (Experimental): Increased intake of whole grain and rye bread
  Interventions: Dietary Supplement: Increased intake of whole grain and rye bread
- C (Active Comparator): Control diet with decreased intake of rye bread, berries and fish
  Interventions: Dietary Supplement: Control diet with decreased intake of rye bread, berries and fish

INTERVENTIONS:
Dietary Supplement: Diet with increased intake of rye bread, berries and fish — Dietary modification with commercial food items
  Arms: A
Dietary Supplement: Increased intake of whole grain and rye bread — Dietary modification with commercial food items
  Arms: B
Dietary Supplement: Control diet with decreased intake of rye bread, berries and fish — Dietary modification with commercial food items
  Arms: C

SUMMARY:
Professor Matti Uusitupa, University of Kuopio, Department of Clinical Nutrition (www.uku.fi) Docent Matej Oresic, VTT (www.vtt.fi) Ursula Schwab, PhD, Docent, Marjukka Kolehmainen, PhD, Docent, Leena Pulkkinen, PhD, Docent, David Laaksonen, MD, PhD, MPH, Docent, Kaisa Poutanen, DSc (Tech), Research Professor

ABSTRACT

The metabolic syndrome (MS) and type 2 diabetes (T2DM) are the most important health problems worldwide. In Finland the prevalence of T2DM is 12-15% among middle-aged people. The prevalence of less marked disturbances in glucose metabolism and MS is 30-40%. Because MS and T2DM are important risk factors for cardiovascular diseases (CVD), the leading cause of death in western countries, all efforts to reverse the epidemic increase in the incidence of MS and T2DM are warranted. The investigators have focused for years on the prevention and non-pharmacological treatment of T2DM and its complications including studies on genetic regulation of glucose and lipid metabolism after dietary modifications. In the investigators' recent projects, the investigators have studied the effects of long-term dietary interventions on gene expression profiles of fat tissue in subjects who are at risk of T2DM. The ultimate goal of these projects has been to identify genes and gene clusters and their biological pathways that respond to dietary modification and modulate glucose and lipid metabolism, and to develop dietary strategies for prevention of T2DM. The main goal of this project is to find nutrition related early biomarkers for progression of MS to T2DM by using modern technologies of systems biology (transcriptomics, metabolomics) of carefully conducted dietary interventions involving subjects with MS. The data will be analysed by using bioinformatics. The investigators reflect these new data to well-known risk factors for T2DM and CVD, e.g., insulin sensitivity, insulin secretion, serum lipids and inflammatory factors among others. In addition to interventions conducted earlier, a new intervention with a whole grain-berry-fish diet and a whole grain diet compared to a control diet with refined foods will be performed. The aim is to increase the investigators' understanding on the synergistic effects of these foods, because the investigators' previous interventions have shown that these individual foods have beneficial effects on glucose and lipid metabolism. On the contrary, diets with refined foods may be harmful in long-term due to its high insulin response, which may through chronic stress lead to both insulin resistance and beta-cell damage.

The significance of this project is to increase understanding of the pathophysiology of MS, T2DM and CVD in physiological, cellular and genetic systems, which may lead to more effective and individualised strategies for treatment and prevention, and better identification of high-risk individuals responsive to specific dietary modifications. Increasing knowledge of dietary factors involved in the progression of MS to T2DM and CVD offers new opportunities to individually tailored diets in the management and prevention of these disorders. The results will also be beneficial for the food industry in developing new functional foods. These results and actions may help delay or even stop the epidemic of MS and T2DM and their negative effect on public health currently seen in Finland and worldwide.

ELIGIBILITY:
Inclusion Criteria:

* impaired glucose tolerance (oral glucose tolerance test with 2-h glucose concentration 7,8-11,0 mmol/l) OR
* impaired fasting glucose fasting plasma glucose concentration 5,6-6,9 mmol/l = IFG)
* and two of the criteria for metabolic syndrome:
* BMI 26-39 kg/m2
* Waist circumference > 102 cm (men) or > 88 cm (women)
* hypertriglyceridemia (fasting serum triglyceride conc > 1,7 mmol/l),
* HDL-cholesterol (fasting serum HDL conc < 1,0 mmol/l for men and < 1,3 mmol/l for women)
* Blood pressure ≥ 130/≥ 85 mmHg

Exclusion Criteria:

* BMI > 40 kg/m2
* fasting serum triglyceride conc > 3.5 mmol/l
* fasting serum cholesterol > 8 mmol/l
* type 1 or 2 diabetes
* abnormal liver, kidney or thyroid function
* large alcohol intake (women >16, men > 24 doses (4cl liquor or equivalent) during week)
* inflammatory bowel disease
* disease that prevents participation
* neuroleptic neuroleptic cortisone medication

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2007-09; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Changes in glucose metabolism, changes in transcriptomic and metabolomic profiles | By 2010

SECONDARY OUTCOMES:
Interaction between the diet and genetic factors within treatment groups | By 2010

CONTACTS AND LOCATIONS:
Overall Officials: Matti IJ Uusitupa, professor, rector, Study Director — University of Kuopio, Department of Clinical Nutrition
Locations (1):
- University of Kuopio, Department of Clinical Nutrition, Kuopio, Finland

REFERENCES:
- [Derived] Karkkainen O, Lankinen MA, Vitale M, Jokkala J, Leppanen J, Koistinen V, Lehtonen M, Giacco R, Rosa-Sibakov N, Micard V, Rivellese AAA, Schwab U, Mykkanen H, Uusitupa M, Kolehmainen M, Riccardi G, Poutanen K, Auriola S, Hanhineva K. Diets rich in whole grains increase betainized compounds associated with glucose metabolism. Am J Clin Nutr. 2018 Nov 1;108(5):971-979. doi: 10.1093/ajcn/nqy169. PMID 30256894
- [Derived] Lankinen MA, Hanhineva K, Kolehmainen M, Lehtonen M, Auriola S, Mykkanen H, Poutanen K, Schwab U, Uusitupa M. CMPF does not associate with impaired glucose metabolism in individuals with features of metabolic syndrome. PLoS One. 2015 Apr 15;10(4):e0124379. doi: 10.1371/journal.pone.0124379. eCollection 2015. PMID 25874636
- [Derived] Hanhineva K, Lankinen MA, Pedret A, Schwab U, Kolehmainen M, Paananen J, de Mello V, Sola R, Lehtonen M, Poutanen K, Uusitupa M, Mykkanen H. Nontargeted metabolite profiling discriminates diet-specific biomarkers for consumption of whole grains, fatty fish, and bilberries in a randomized controlled trial. J Nutr. 2015 Jan;145(1):7-17. doi: 10.3945/jn.114.196840. Epub 2014 Nov 12. PMID 25527657
- [Derived] Lankinen M, Kolehmainen M, Jaaskelainen T, Paananen J, Joukamo L, Kangas AJ, Soininen P, Poutanen K, Mykkanen H, Gylling H, Oresic M, Jauhiainen M, Ala-Korpela M, Uusitupa M, Schwab U. Effects of whole grain, fish and bilberries on serum metabolic profile and lipid transfer protein activities: a randomized trial (Sysdimet). PLoS One. 2014 Feb 28;9(2):e90352. doi: 10.1371/journal.pone.0090352. eCollection 2014. PMID 24587337
- [Derived] Lappi J, Salojarvi J, Kolehmainen M, Mykkanen H, Poutanen K, de Vos WM, Salonen A. Intake of whole-grain and fiber-rich rye bread versus refined wheat bread does not differentiate intestinal microbiota composition in Finnish adults with metabolic syndrome. J Nutr. 2013 May;143(5):648-55. doi: 10.3945/jn.112.172668. Epub 2013 Mar 20. PMID 23514765
- [Derived] Lankinen M, Schwab U, Kolehmainen M, Paananen J, Poutanen K, Mykkanen H, Seppanen-Laakso T, Gylling H, Uusitupa M, Oresic M. Whole grain products, fish and bilberries alter glucose and lipid metabolism in a randomized, controlled trial: the Sysdimet study. PLoS One. 2011;6(8):e22646. doi: 10.1371/journal.pone.0022646. Epub 2011 Aug 25. PMID 21901116
- [Derived] de Mello VD, Schwab U, Kolehmainen M, Koenig W, Siloaho M, Poutanen K, Mykkanen H, Uusitupa M. A diet high in fatty fish, bilberries and wholegrain products improves markers of endothelial function and inflammation in individuals with impaired glucose metabolism in a randomised controlled trial: the Sysdimet study. Diabetologia. 2011 Nov;54(11):2755-67. doi: 10.1007/s00125-011-2285-3. Epub 2011 Aug 26. PMID 21870174